CLINICAL TRIAL: NCT05580081
Title: Optimizing CBT Implementation Among Community Providers Through Internet-based Consultation and Networking (i-CAN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A22-0473
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; CBT
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The RCT is a parallel group design, in which those in Control will be offered i-CAN after the 18 week waiting period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-CAN (Experimental): 18 weeks of access to the online consulting platform
  Interventions: Behavioral: i-CAN
- waitlist control (No Intervention): No offered support or consultation

INTERVENTIONS:
Behavioral: i-CAN — online support and consultation to providers
  Arms: i-CAN

SUMMARY:
Although anxiety is one of the most common and debilitating mental health conditions affecting children and adolescents, the vast majority of sufferers do not receive effective treatment. Cognitive-behavioral therapy (CBT) is an evidence-based, frontline treatment for pediatric anxiety, yet many community-based practitioners do not implement CBT with high fidelity, which can detrimentally affect its clinical impact. The goal of this study is to develop and test an online platform to support community providers' effective use of CBT for pediatric anxiety.

DETAILED DESCRIPTION:
Stemming from implementation science and, specifically, the Theory of Planned Behavior, investigators are working alongside community stakeholders to develop a novel, online consultation platform. This platform, termed Internet-based Consultation or Networking (or i-CAN) will utilize a professional navigator (i.e., a provider with CBT expertise), online support and resources, and parallel peer consultation to create a user-friendly and supportive community for providers to get support as they implement CBT. Once finalized, the platform will be tested in the context of a preliminary randomized controlled trial (RCT) with approximately 100 mental healthcare providers who work with anxious children and adolescents. Providers who enroll will be randomly assigned to either the experimental condition (i-CAN) or the control condition (wait-list for i-CAN). The primary outcome of interest is change in intentions to use CBT.

ELIGIBILITY:
Inclusion Criteria:

* provide direct mental healthcare to anxious youth
* practice in general community within state of Alabama
* agree to try i-CAN

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Reasoned Action Questionnaire | 18 weeks
  Questionnaire that assesses instrumental beliefs, perceived norms, and self-efficacy (all related to use of cognitive-behavioral therapy). On the Reasoned Action Questionnaire, higher scores indicate greater intention to use the therapeutic approach. Scores can range from 14 to 90.

SECONDARY OUTCOMES:
Evidence-based practice attitude scale | 18 weeks
  Questionnaire that assesses views toward cognitive-behavioral therapy. Higher scores indicate more positive views. Scores can range from 0 to 60.

CONTACTS AND LOCATIONS:
Overall Officials: Susan W White, PhD, Principal Investigator — UA
Locations (1):
- Center for Youth Development and Intervention, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared to NDA, and data requests can be issued directly to NDA.